CLINICAL TRIAL: NCT05966610
Title: Bizarreness and Anomalous Self Experiences in Schizophrenia: Pilot Study on Diagnostic Decision-Making
Brief Title: Bizarreness and Anomalous Self Experiences in Schizophrenia
Acronym: BASES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0517; 2023-A00049-36 (Other: ID-RCB)
Record Dates: First submitted 2023-05-30; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: Praecox Feeling; Self-Disorders; Subjectivity; Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several authors suggest that the specific experience felt in clinical encounter, called Praecox Feeling, is directly linked to the psychopathology of Schizophrenia.

However, determining factors of this phenomena, whether cognitive or subjective, remains poorly studied.

Furthermore, Self-Disorders are alterations of the first-person experience regarded as specific of the disease. The investigators plan to study in an exploratory way the phenomenological and subjective links between Praecox Feeling and Self Disorders determinants, while hypothesizing that the clinician's Praecox Feeling can be positively correlated to SDs, as our main objective.

DETAILED DESCRIPTION:
Several authors suggest that the specific experience felt in clinical encounter, called Praecox Feeling, is directly linked to the psychopathology of Schizophrenia. However, subjective, cognitive or neurophysiologic aspects of this phenomena remains poorly studied.

Furthermore, Self-Disorders (SD) are alterations of the first-person experience and of sense of agency, regarded as specific of Schizophrenia. Unlike Praecox Feeling, clinical, cognitive and neuropsychological determinants of SD are increasingly studied.

The investigators plan to study in an exploratory way the links between Praecox Feeling and SDs determinants, while hypothesizing that the clinician's Praecox Feeling can be positively correlated to SDs, as our main objective.

As a secondary outcome, the investigators will control this correlation by a comparison between SDs evaluation and clinician subjectivity.

The present study also plan to evaluate the associations between Praecox Feeling and clinical features, low and high cognitive level with attentional and social cognition evaluations.

The first step of the research project is to implement this exploratory design in a transversal multicentric setting between centers with a limited number of participants and without follow-up.

ELIGIBILITY:
Inclusion Criteria:

* People with a diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria.
* Psychiatric medical situation judged clinically stable : no change of main antipsychotic in treatment in last 15 days.
* People who has given his non-opposition
* Patients affiliated to a social security system

Exclusion Criteria:

* Previous meeting of the participant with one of the investigators involved in the clinical assessment and scoring of the study scales.
* Person with a moderate to severe intellectual disability (clinical criteria).
* Person with a neurological pathology with cognitive impact
* Patients with legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stabilised patients with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between Praecox Feeling and Self Disorders | 2 months
  Comparison between Examination of Anomalous Subjective Experience (EASE) total score evaluated at third visit and mean of Praecox Feeling intensity measured by a visual analog scale (VAS) evaluated at each visit.
  Examination of Anomalous Subjective Experience is a 5-item interview asked by the investigator.
  Visual Analog Scale (VAS) is a scale that evaluates the level of strangeness felt during the patient/investigator encounter. It goes from 0 (no strangeness feeling) to 100 (maximal strangeness feeling).

SECONDARY OUTCOMES:
Correlation between Praecox Feeling and symptomatic dimensions | 2 months
  Comparison between mean of Praecox Feeling intensity measured by a visual analog scale evaluated at each visit and Cognition evaluation in second visit with attentional evaluation (D2-R and results at Go/No-Go testing) and social cognition evaluation (TOM-15).
  D2-R is a paper-and-pencil test. It's consists of the subject identifying and crossing out target characters (d with 2 lines) from a large number of characters.
  Go/No-Go testing is a test assesses behavioural control in a test where the participant must be able to respond to an automated external stimulus.
  TOM-15 consists of a false belief task and a comprehension task using the same 15 stories but different questions. The stories proposed show everyday situations. There are 8 first-order questions and 7 second-order questions, allowing two scores to be calculated, one for each order (maximum 15 in total). The more correct answers, the higher the score
Correlation between Praecox Feeling intensity and Self Disorders intensity | 2 months
  Comparison between Examination of Anomalous Subjective Experience (EASE) total score a the third visit and mean of clinician subjectivity measured by Assessment of clinician's subjective experience (ACSE) at each visit.
  Examination of Anomalous Subjective Experience is a scale completed during the clinical interview by the investigator. It consists a 5-item scale.
  Assessment of clinician's subjective experience is a scale completed during the clinical interview by the investigator. It is composed of 45 items.
Correlation between the patient's judgment and the quality of the meeting | 2 months
  Meeting Quality, according to the participant, evaluated at second visit in an unstructured way.

CONTACTS AND LOCATIONS:
Overall Officials: Tudi GOZE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France